CLINICAL TRIAL: NCT07402694
Title: Oral Health Outcomes With Amphion Mouthwash as an Adjunct to Non-Surgical Periodontal Therapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-2053
Record Dates: First submitted 2026-01-11; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Mouthwash
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amphion® Mouthwash Group (Experimental): Receives non-surgical periodontal therapy followed by irrigation and daily rinsing with Amphion® Mouthwash containing the active ingredient.
  Interventions: Drug: Amphion® Mouthwash
- Placebo Mouthwash Group (Placebo Comparator): Receives non-surgical periodontal therapy followed by irrigation and daily rinsing with a placebo mouthwash identical in appearance, odor, and taste but containing no active ingredient.
  Interventions: Drug: Placebo Mouthwash

INTERVENTIONS:
Drug: Amphion® Mouthwash — All enrolled subjects first receive non-surgical periodontal treatments (scaling, root planing, debridement). Upon completion, they immediately undergo periodontal irrigation with Amphion® Mouthwash according to their group assignment and receive standardized oral hygiene instructions. Subsequently, subjects begin the home rinsing regimen: twice daily (morning and evening), using 15 mL of Amphion® Mouthwash for 1 minute per rinse before expectorating.
  Arms: Amphion® Mouthwash Group
Drug: Placebo Mouthwash — All enrolled subjects first receive non-surgical periodontal treatments (scaling, root planing, debridement). Upon completion, they immediately undergo periodontal irrigation with Placebo Mouthwash according to their group assignment and receive standardized oral hygiene instructions. Subsequently, subjects begin the home rinsing regimen: twice daily (morning and evening), using 15 mL of Placebo Mouthwash for 1 minute per rinse before expectorating.
  Arms: Placebo Mouthwash Group

SUMMARY:
Periodontitis is a chronic inflammation caused by dental plaque that can destroy periodontal tissues. Current primary treatments include mechanical removal methods such as supragingival scaling and subgingival curettage. However, issues like microbial recolonization leading to inflammation recurrence exist, often necessitating the use of antimicrobial agents. Prolonged antibiotic use, however, can easily lead to bacterial resistance.

Amphion oral rinse is a novel biomimetic material mouthwash. It inhibits plaque regrowth by forming a long-lasting physical barrier and avoids flora imbalance. Compared with traditional antibiotics, this product has shown unique advantages in the adjuvant treatment of periodontal diseases. This study aims to evaluate the efficacy of Amphion rinse combined with conventional periodontal therapy in patients with stage I-IV periodontitis, including plaque control and inflammation improvement. Additionally, it will analyze its impact on the oral microbiome and collect user experience feedback to provide a reference for its clinical application.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease initiated by dental plaque biofilm as the primary etiological factor. Its main pathological feature is the progressive destruction of periodontal supporting tissues. Currently, mechanical removal of dental calculus and plaque remains the foundational treatment for periodontitis, primarily consisting of supragingival scaling, subgingival curettage, and root planing. However, such treatments have certain limitations: microorganisms from other areas in the oral cavity can recolonize the periodontal pockets, leading to disease recurrence. Therefore, the adjuvant use of antimicrobial agents is often necessary. Nevertheless, long-term or extensive use of antibiotics can easily induce bacterial resistance, resulting in the gradual evolution of various pathogenic bacteria associated with human diseases into multidrug-resistant strains.

Amphion oral rinse is a mouthwash developed based on cell membrane-mimicking polymer materials, with its core breakthrough being its "zero immunogenicity" property. By forming a long-lasting physical barrier on the oral surface, this product effectively inhibits plaque regrowth and avoids side effects such as flora imbalance caused by broad-spectrum antimicrobial activity. The duration of its barrier effect can exceed 7 days. Consequently, in the treatment of periodontal diseases, Amphion oral rinse demonstrates potential advantages over traditional antibiotic-based medications. It is expected to serve as an effective means of plaque control, complementing mechanical therapies and other approaches to eliminate periodontal pathogenic microorganisms, reduce or eliminate local inflammatory responses, and thereby achieve the goal of adjuvant treatment for periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 years old.
2. At least 20 natural teeth (excluding root remnants) present in the oral cavity.
3. Diagnosed with Stage I-IV periodontitis according to the 2018 new classification of periodontal diseases.
4. No impairment in vision, motor function, or cognitive ability, capable of understanding and cooperating with the study.
5. Not undergoing any orthodontic treatment and not wearing removable partial dentures during the study period.
6. Fully informed and voluntarily signed a written informed consent form.

Exclusion Criteria:

1. Individuals allergic to any component used in the study.
2. Pregnant or lactating women.
3. Those who have undergone periodontal treatments such as scaling, root planing, or used antimicrobial mouthwash within the past 3 months.
4. Those with a history of systemic hormone or antibiotic use within the past 3 months, or who are assessed as requiring adjunctive use of such medications during periodontal treatment.
5. Individuals with underlying systemic diseases that may affect the evaluation of periodontal status, including but not limited to: abnormal liver function, renal insufficiency, hematological diseases, neurological or psychiatric disorders, systemic bone diseases, diabetes, coronary heart disease, malignant tumors, etc.
6. Current or former smokers (including active or passive smoking), or users of other nicotine and tobacco products (such as e-cigarettes, chewing tobacco).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean full-mouth Plaque Index (PI) | Before treatment (baseline), and at 6 weeks and 3 months after treatment.
  The PI assesses the thickness of plaque at the gingival margin. Four sites per tooth (mesial, distal, buccal, lingual) are scored from 0 (no plaque) to 3 (abundance of plaque). A lower score indicates better oral hygiene. The outcome will be reported as the mean PI score per patient across all examined sites.

SECONDARY OUTCOMES:
Mean full-mouth Bleeding Index (BI) | Pre-treatment (baseline), 6 weeks post-treatment, and 3 months post-treatment
  The BI assesses gingival inflammation by recording bleeding upon gentle probing. Each tooth is probed at four sites (mesial, distal, buccal, lingual) and scored as 0 (no bleeding within 30 seconds) or 1 (bleeding present). A lower score indicates healthier gingiva. The outcome will be reported as the mean BI score per patient (percentage of bleeding sites).
Mean Pocket Probing Depth (PPD) | Pre-treatment (baseline), 6 weeks post-treatment, and 3 months post-treatment
  PPD is measured from the gingival margin to the base of the pocket using a periodontal probe. Measurements will be taken at six sites per tooth (mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual, distolingual). The outcome will be reported as the mean PPD in millimeters per patient for all measured sites.
Mean Clinical Attachment Level (CAL) | Pre-treatment (baseline), 6 weeks post-treatment, and 3 months post-treatment
  CAL is the distance from the Cemento-Enamel Junction (CEJ) to the base of the pocket, measured with a periodontal probe. It indicates the historical loss of periodontal support. Measurements at six sites per tooth. The outcome will be reported as the mean CAL in millimeters per patient for all measured sites.
Microbial composition of subgingival plaque (relative abundance of key periodontal pathogens) | Pre-treatment (baseline), 6 weeks post-treatment, and 3 months post-treatment
  Subgingival plaque samples will be collected from pre-selected deep pockets. Microbial composition (e.g., relative abundance of Porphyromonas gingivalis, Treponema denticola, Tannerella forsythia) will be analyzed via 16S rRNA gene sequencing or specific PCR. The outcome will be reported as the change in relative abundance (%) of target pathogens from baseline.
Microbial composition of salivary plaque (total bacterial load and diversity) | Baseline (pre-treatment), 6 weeks, and 3 months post-treatment
  Unstimulated whole saliva will be collected. Total bacterial load (by quantitative PCR) and microbial alpha-diversity (e.g., Shannon Index) will be assessed. The outcome will be reported as the change in total bacterial count (gene copies/mL) and Shannon Index value from baseline.
Root surface hypersensitivity assessed by a Visual Analogue Scale (VAS) | Pre-treatment (baseline), 6 weeks post-treatment, and 3 months post-treatment
  Participants rate their level of tooth sensitivity to cold air/water on a 100-mm horizontal VAS, where 0 mm = "No pain" and 100 mm = "Unbearable pain". A lower score indicates less sensitivity. The outcome will be reported as the mean VAS score (mm) per patient.
Alteration in taste sensation assessed by a 5-point Likert scale | 6 weeks and 3 months post-treatment (during rinsing period).
  Participants report any change in taste sensation using a questionnaire with a Likert scale from 1 (Much Worse) to 5 (Much Better). A score of 3 indicates "No Change". The outcome will be reported as the frequency and percentage of patients in each response category.
Patient adherence to rinsing regimen (days of rinsing completed) | Through study completion, an average of 6 weeks
  Adherence is monitored via patient diary and bottle return/weighing. The outcome will be reported as the percentage of prescribed rinsing days completed (e.g., 90% adherence means the subject performed rinsing on 81 out of 90 expected days).
Periodontitis Staging and Grading | Baseline.
  The specific stage (I, II, III, IV, reflecting disease severity and complexity) and grade (A, B, C, reflecting the rate of progression and risk assessment) of periodontitis will be recorded for each patient according to the 2018 new classification of periodontal diseases. This will serve as a key baseline variable for subgroup analysis.
Medication History | Baseline
  A systematic record of the patient's current long-term medication use, particularly drugs that may affect periodontal tissues or healing (e.g., calcium channel blockers, anticonvulsants, immunosuppressants, long-term NSAIDs, etc.). Categorized as "Yes" or "No".
Oral Health-Related Quality of Life (OHRQoL) | Baseline, 3 months post-treatment
  Assessment using a validated short-form scale (e.g., Oral Health Impact Profile-14, OHIP-14). The scale contains 14 questions covering dimensions such as functional limitation, pain, and psychological discomfort. A higher total score indicates a greater negative impact of oral health on quality of life.
Age | Baseline
  Age in years at the time of enrollment.
Gender | Baseline
  Self-reported gender, categorized as Male or Female.
Body Mass Index (BMI) | Baseline.
  Body mass index calculated as weight in kilograms divided by height in meters squared (kg/m²). Categorized per Chinese Adult Guidelines: Underweight (<18.5 kg/m²), Normal (18.5-23.9 kg/m²), Overweight (24.0-27.9 kg/m²), Obese (≥28.0 kg/m²).
Tooth Brushing - Frequency | Before treatment (baseline), and at 6 weeks and 3 months after treatment.
  Self-reported frequency of daily tooth brushing. Categorized as: Once per day, Twice per day, More than twice per day, or Occasionally/Not every day.
Tooth Brushing - Method | Before treatment (baseline), and at 6 weeks and 3 months after treatment.
  Self-reported primary tooth brushing technique (e.g., Horizontal scrub, Bass method, Vertical sweep, etc.).
Tooth Brushing - Duration | Before treatment (baseline), and at 6 weeks and 3 months after treatment.
  Self-reported average time spent brushing per session, in seconds/minutes. Categorized (e.g., <1 minute, 1-2 minutes, >2 minutes).
Use of Dental Floss/Interdental Cleaners | Before treatment (baseline), and at 6 weeks and 3 months after treatment.
  Self-reported use of interdental cleaning aids. Assessed by type (dental floss, interdental brush) and frequency (e.g., Daily, Several times per week, Occasionally, Never).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu J, Huang Y, Lou X, Liu B, Liu W, An N, Wu R, Ouyang X. Effect of Pudilan Keyanning antibacterial mouthwash on dental plaque and gingival inflammation in patients during periodontal maintenance phase: study protocol for double-blind, randomised clinical trial. BMJ Open. 2021 Nov 2;11(11):e048992. doi: 10.1136/bmjopen-2021-048992. PMID 34728444
- [Result] Nardi GM, Cesarano F, Papa G, Chiavistelli L, Ardan R, Jedlinski M, Mazur M, Grassi R, Grassi FR. Evaluation of Salivary Matrix Metalloproteinase (MMP-8) in Periodontal Patients Undergoing Non-Surgical Periodontal Therapy and Mouthwash Based on Ozonated Olive Oil: A Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Sep 11;17(18):6619. doi: 10.3390/ijerph17186619. PMID 32932898
- [Result] Shaheen MY, Al-Zawawi AS, Divakar DD, Aldulaijan HA, Basudan AM. Role of Chlorhexidine and Herbal Oral Rinses in Managing Periodontitis. Int Dent J. 2023 Apr;73(2):235-242. doi: 10.1016/j.identj.2022.06.027. Epub 2022 Jul 28. PMID 35907673
- [Result] Rath A, Wong M, Li K, Wong A, Tan L, Tan K, Pannuti CM. Efficacy of adjunctive octenidine hydrochloride as compared to chlorhexidine and placebo as adjuncts to instrumentation in stage I-II periodontitis: A double-blinded randomized controlled trial. Int J Dent Hyg. 2024 Nov;22(4):802-813. doi: 10.1111/idh.12795. Epub 2024 Mar 10. PMID 38461488
- [Result] Sparabombe S, Monterubbianesi R, Tosco V, Orilisi G, Hosein A, Ferrante L, Putignano A, Orsini G. Efficacy of an All-Natural Polyherbal Mouthwash in Patients With Periodontitis: A Single-Blind Randomized Controlled Trial. Front Physiol. 2019 May 22;10:632. doi: 10.3389/fphys.2019.00632. eCollection 2019. PMID 31191341
- [Result] Matayoshi S, Tojo F, Suehiro Y, Okuda M, Takagi M, Ochiai M, Kadono M, Mikasa Y, Okawa R, Nomura R, Itoh Y, Itoh N, Nakano K. Effects of mouthwash on periodontal pathogens and glycemic control in patients with type 2 diabetes mellitus. Sci Rep. 2024 Feb 2;14(1):2777. doi: 10.1038/s41598-024-53213-x. PMID 38307981
- [Result] Waqar SM, Razi A, Qureshi SS, Saher F, Zaidi SJA, Kumar C. Comparative evaluation of propolis mouthwash with 0.2% chlorhexidine mouthwash as an adjunct to mechanical therapy in improving the periodontitis among perimenopausal women: a randomized controlled trial. BMC Oral Health. 2024 Jan 5;24(1):26. doi: 10.1186/s12903-023-03768-4. PMID 38183081
- [Result] Ozmeric N, Enver A, Isler SC, Gokmenoglu C, Topaloglu M, Selamet H, Altun G, Aykol Sayar S. Evaluating the effects of chlorhexidine and vitamin c mouthwash on oral health in non-surgical periodontal therapy: a randomized controlled clinical trial. Sci Rep. 2025 Jan 29;15(1):3703. doi: 10.1038/s41598-025-88100-6. PMID 39881161
- [Result] Teng F, He T, Huang S, Bo CP, Li Z, Chang JL, Liu JQ, Charbonneau D, Xu J, Li R, Ling JQ. Cetylpyridinium chloride mouth rinses alleviate experimental gingivitis by inhibiting dental plaque maturation. Int J Oral Sci. 2016 Sep 29;8(3):182-90. doi: 10.1038/ijos.2016.18. PMID 27680288